CLINICAL TRIAL: NCT06725654
Title: Evaluation of Oral and Dental Health of Institutionalized Orphan Children Residing in Children's Homes in Turkey
Status: Completed | Type: Observational
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Arzu Koçkanat, Assistant Professor, Cumhuriyet University
Other Study IDs: CumhuriyetU_ArzuKockanat_001
Record Dates: First submitted 2024-12-02; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Dental Caries; Orphaned Children; Periodontal Index
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Institutionalized Orphan Children Residing in Children's Homes: Institutionalized orphan children reside in children's homes in Sivas, Turkey.
  Interventions: Other: Diagnostic Procedures

INTERVENTIONS:
Other: Diagnostic Procedures — To evaluation the oral and dental health of orphaned children, DMFT, deft, GI, PI and CPITN indices were used to assess dental caries experience, gingival inflammation, the amount of plaque on the tooth surface and periodontal status, respectively.

SUMMARY:
Both dental caries prevalence and periodontal status of children residing in children's homes in Sivas province of Turkey were evaluated.

DETAILED DESCRIPTION:
This study was carried out in 16 state-protected children's homes in Sivas under the Directorate of Coordination of Children's Homes Centres of the Ministry of Family and Social Policies of Turkey. A total of institutionalized 90 orphan children between the ages of 6 and 18, who did not have any chronic diseases, were not taking medication, and were compliant and healthy, were included in the study. Since all participants of this study are under state protection, Sivas Children's Homes Center Coordination Directorate was contacted. The aim of the study and the procedures were explained in detail and official permission was obtained. The children's caregivers signed informed consent forms approved by the Ethics Committee. The examination procedures were performed by two trained dentists as recommended by the WHO. DMFT and deft, GI and PI indices were used to assess dental caries experience, gingival inflammation, and the amount of plaque on the tooth surface, respectively. Also, periodontal status and treatment need were evaluated using the CPITN index.

ELIGIBILITY:
Inclusion Criteria:

* Does not have any chronic disease.
* Not taking any medication.
* To be compatible and healthy.

Exclusion Criteria:

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Orphaned children aged from 6 to 18 years old residing in children's home who meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Caries Experience | Immediately after the orphans filled the survey forms at the first visit
  Oral and dental examination was done by a specialist pedodontist, and DMFT index (total number of decayed, filled, and missing teeth) was recorded.
Gingival Index (GI, Löe and Sillness-1963) measurements | Immediately after the orphans filled the survey forms at the first visit
  In order to determine the gingival inflammation of the participants, the Löe & Silness gingival index values (GI) were evaluated by a specialist periodontist by scoring the mesial, distal, lingual and vestibular gingival conditions of the teeth (16, 11, 24, 31, 36, 44) determined in each sextant between 0 and 3 (Score 0: healthy gingiva, no inflammation, Score 1: mild inflammation, discoloration and mild edema in the gingiva, no bleeding on probing, Score 2: moderate inflammation, redness and edema in the gingiva, bleeding on probing, Score 3: severe inflammation, redness and edema in the gingiva, spontaneous bleeding).
Plaque Index (PI, Sillness and Löe-1964) measurements | Immediately after the orphans filled the survey forms at the first visit
  In order to determine the amount of plaque on the tooth surface of the participants, Silness & Löe plaque index values (PI) were evaluated by a specialist periodontist by scoring the mesial, distal, lingual and vestibule gingival conditions of the teeth (16, 11, 24, 31, 36, 44) determined in each sextant between 0 and 3.(Score 0: No bacterial plaque on the tooth surface. Score 1:There is plaque in the form of film and can be seen with the help of a probe. Score 2:There is moderate soft attachment visible to the naked eye. Score 3:There is a visible dense soft appendage filling the gingival sulcus on the tooth surface.)
Community Periodontal Index of Treatment Needs (CPITN) | Immediately after the orphans filled the survey forms at the first visit
  CPI values used to determine the need for community periodontal treatment were determined by a specialist periodontist by scoring between 0 and 4 (Score 0: healthy periodontium, Score 1: bleeding after probing, no calculus/iatrogenic irritation, Score 2: presence of supra and/or subgingival calculus, presence of iatrogenic perforation, Score 3: presence of shallow pockets between 3.5 and 5.5 mm, Score 4: presence of pockets deeper than 5.5 mm). The following scores were used to determine the TN values. (Score 0: No need additional treatment, Score 1: oral hygiene instruction improvement in personal oral hygiene, Score 2: scaling oral hygiene instruction, Score 3: periodontal treatment infected tissue, Score 4: complex periodontal treatment.)

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Koçkanat, Asst.Prof., Principal Investigator — Cumhuriyet University
Locations (1):
- Cumhuriyet University, Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kockanat A, Acipinar S. Evaluation of oral and dental health of institutionalized orphan children residing in children's homes in Turkiye. BMC Oral Health. 2025 Nov 24;25(1):1829. doi: 10.1186/s12903-025-07240-3. PMID 41286857